CLINICAL TRIAL: NCT06116279
Title: First-in-human Experience Using Novel Ultraflexible Low-impedance Electrode Arrays: an IDEAL Stage 1 Study
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Great Ormond Street Hospital for Children NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 21BI27
Record Dates: First submitted 2023-07-26; First posted 2023-11-03 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Epilepsy; Focal Cortical Dysplasia
Keywords: Epilepsy; FCD; LEAT; Neurosurgery; Microelectrode; Local field potential; Epileptic zone
MeSH Terms: conditions — Epilepsy; Focal Cortical Dysplasia

STUDY DESIGN:
Intervention Model Description: The investigators will adhere to the internationally accepted five-stage Idea, Development, Evaluation, Assessment, Long-term study (IDEAL) framework for novel surgical device innovation. An IDEAL Stage 1 study requires a highly-selected patient group (n=6) and focuses on novel device innovation feasibility and safety. Adhering to the IDEAL framework will facilitate the development and evaluation of the novel device in a logical manner that balances innovation and safety.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Insertion of electrode during planned neurosurgery for epilepsy (Experimental): During the surgical procedure, following exposure of the brain via a craniotomy, the novel electrodes will be inserted into tissue planned for resection. This will be targeted using the existing neuronavigation software that is being used during the surgery and may be augmented by intraoperative ultrasound, also a common adjunct used in these surgeries. Following insertion of the electrode, the cables will be connected to a specialised (portable) amplifier inside the operating theatre and 15 minutes of data will be recoded. The electrodes will then be removed and the surgical resection will then proceed as planned. The content of the recordings will not be available in real-time and will not be used to inform or change the surgical resection plan in any way.
  Interventions: Device: Insertion of electrode during planned neurosurgery for epilepsy

INTERVENTIONS:
Device: Insertion of electrode during planned neurosurgery for epilepsy — A novel, 300 micrometer, ultraflexible, low-impedance electrode proposes to cause minimal parenchymal (brain tissue) damage, and provide multiple contacts at multiple depths to allow unit-level recordings for a period of 15 minutes.

SUMMARY:
The goal of this first-in-human study is to evaluate a novel ultraflexible microelectrode in children undergoing neurosurgery to remove tissue that causes epilepsy (seizures) in focal cortical dysplasia (FCD) or long-term epilepsy-associated tumours (LEAT).

The main questions it aims to answer are:

1. The safety and feasibility of the novel microelectrode into current operative workflow
2. The unique electrophysiological tissue signatures in FCD or LEAT

DETAILED DESCRIPTION:
Epilepsy affects 100,000 people under 25. Many children with epilepsy also have a learning disability or developmental problems and 25-30% continue to have seizures despite best medical treatment.

Neuromodulation or brain stimulation is the delivery of electricity to the brain cells. It may alter the brain activity and overall brain connectivity and currently is rarely used as a treatment for epilepsy. However, it has the potential to reduce the number of seizures and improve other problems that children with epilepsy may have such as concentration, memory and learning. 'Precision neuromodulation', which involves individually tailored treatments requires us to identify where in the brain to stimulate and what the best settings are in each individual. A limitation of current neuromodulation treatment is limited understanding of the abnormal signatures of electrical activity in abnormal tissue.

The investigators have developed a novel electrode that can record signals from the brain at higher resolution than current electrodes. The 2 micrometer, ultraflexible, low-impedance electrode arrays are smaller, less damaging, and provide multiple contacts at multiple depths. The investigators propose a first-in-human study to investigate the feasibility and safety of using these electrodes in patients undergoing surgery for epilepsy - either focal cortical dysplasia (FCD) or long-term associated epilepsy tumours (LEAT).

The investigators will insert the electrode into brain tissue that is going to be removed as part of the planned surgery. The extent of tissue damage caused by insertion will be examined, and whether the electrode is able to capture signals at difference scales from the brain will be assessed; this includes signals from an area of tissue (termed local field potential) and signals from single nerve cells (termed single unit recordings). If safe, it will lay the foundation to use these electrodes in future precision neuromodulation platforms that can be applied to epilepsy and other neurological diseases.

ELIGIBILITY:
Inclusion Criteria:

1. Radiologically visible epileptogenic lesion (focal cortical dysplasia or long-term epilepsy associated tumour) undergoing planned resective surgery

Exclusion Criteria:

1. Unable to provide informed consent

Ages: 3 Months to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 6 (Estimated)
Dates: Start 2024-02-01 (Estimated); Primary Completion 2025-02-01 (Estimated); Study Completion 2025-08-01 (Estimated)

PRIMARY OUTCOMES:
Feasibility of novel electrode into current operative workflow | At operation
  Document total length of set up and recording with electrode (recorded in minutes)

SECONDARY OUTCOMES:
Resected tissue assessed histologically for damage from novel electrode | 4 weeks following operation
  Neuropathologists will perform haematoxylin and eosin histological (H&E), luxol fast blue, and neutral red to describe the insertion tract lesion and neocortical cytoarchitecture
Analysis of recorded electrophysiological data from intraoperative recording by novel electrode | 6 months
  The data obtained from intraoperative recording will be analysed by computational neuroscientists
Safety of novel electrode insertion and recording | At operation
  Intraoperative events occur (haemorrhage, seizure, stroke)

CONTACTS AND LOCATIONS:
Overall Officials: Martin Tisdall, MD FRCS, Principal Investigator — Great Ormond Street Hospital
Locations (1):
- Great Ormond Street Hospital, London, United Kingdom